CLINICAL TRIAL: NCT03329716
Title: A Randomized Controlled Trial Comparing Gradual and Immediate Brace Weaning Protocol
Brief Title: Brace Weaning Protocol Comparing Gradual and Immediate Weaning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Braceweaning001
Record Dates: First submitted 2017-05-02; First posted 2017-11-06 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-05

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: brace weaning

STUDY DESIGN:
Intervention Model Description: A non-blinded, randomized controlled trial for testing two brace weaning protocols, being immediate removal of brace or gradual weaning of brace, over a course of 6 months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Brace Weaning (Other): Immediate weaning of brace
  Interventions: Other: Brace weaning
- Gradual Brace Weaning (Other): Nocturnal brace wearing for 6 months prior to stopping brace
  Interventions: Other: Brace weaning

INTERVENTIONS:
Other: Brace weaning — For AIS patients who have been wearing Boston brace and attend clinic consultation where the decision for brace weaning is made, then weaning protocol of either arm will be prescribed

SUMMARY:
This is a non-blinded, randomized controlled trial for testing two brace weaning protocols namely immediate removal of brace or gradual weaning of brace over a course of 6 months for adolescent idiopathic scoliosis (AIS) patients. These patients will have follow-up visits at 6-months, 12-months and 24-months intervals. By comparing between the two groups in terms of change of Cobb angle, truncal balance, health-related quality of life measures at the set time-points, the investigators aim to gain insights of whether different brace-weaning protocol will be more beneficial in patients' clinical and quality of life measure outcomes.

DETAILED DESCRIPTION:
The aims of this study are: 1) To compare the degree of Cobb angle and truncal balance maintenance between immediate removal and gradual brace weaning protocols for AIS patients who have completed brace treatment; 2) To determine factors for poor maintenance of Cobb angle and truncal balance after brace weaning; 3) To determine if the current standardized criteria for initiating brace weaning is appropriate.

The investigators' hypothesis is that an AIS patient requires gradual brace weaning to allow better adaptation to an unloaded environment without the brace thereby resulting with a better truncal balance. It is also hypothesized that the immediate removal of brace for a AIS patient is as effective in terminating bracing treatment when compared to gradual brace weaning over a 6-month period.

The investigators will recruit AIS patients managed at the Duchess of Kent Children's Hospital (DKCH) in Hong Kong. As there is no definition for "brace weaning", we adopt the protocol that our center has been using. Hence the investigators will be comparing two protocols: 1) brace wearing time shortened to night wearing for 6 more months before stopping bracing altogether or 2) immediate brace weaning on the day of patient recruitment. All patients will be recruited on the day of clinic consultation where the decision for brace weaning is made. Those with underarm (Boston) bracing are included in the study. All subjects are followed-up longitudinally up to 2 years after brace weaning has been issued. Hence this includes three clinic visits with one at 6 months to complete the gradual brace weaning protocol, and at 1 and 2 years to observe for any delayed changes to the overall curvature and balance including loss of truncal balance and Cobb angle deterioration. This does not deviate significantly from our usual care as all AIS subjects are usually followed-up at 6-monthly intervals and thus this duration of follow-up is strictly adherent to and standardized.

Eligible patients who have consented to take part will be randomly allocated to one of the two protocols, and group designation will be decided by a computer-generated randomized table. Restricted randomization through blocking will be used according to the equal proportion rule (1:1). The random allocation sequence will be managed independently, and the random coding is concealed to all research staff until all data analyses have been completed. The clinicians and research assistants will not be blinded to treatment allocation, as the participants are required to implement bracing protocols and schedule longitudinal follow-up.

Apart from the Cobb angle measurement, all subjects undergo weight, height and arm span measurements, health-related quality of life (HRQOL) and utility measurements, and whole spine standing posteroanterior (PA) and lateral radiographs at each clinic visit as per routine clinic protocol. The refined Scoliosis Research Society 22-item (SRS-22r) questionnaire and the EuroQoL 5-Dimension 5-Level (EQ5D) questionnaire will thus be provided at every visit.

ELIGIBILITY:
Inclusion Criteria:

* AIS patients who have been wearing underarm (Boston) bracing, and who have reached skeletal maturity based on the Scoliosis Research Society (SRS) standardized criteria: Risser stage ≥4, >2 years post-menarche, and no growth between 2 visits. The subjects should be managed at the Duchess of Kent Children's Hospital (DKCH) in Hong Kong.

Exclusion Criteria:

* All patients that are not AIS, using Milwaukee bracing, unable to comply with study follow-up, protocol issued and refused consent for study

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 369 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change of Cobb Angle | Baseline, then 6-months, 12-months and 24-months follow-ups
  Cobb angle changes between baseline (when decision to initiate brace weaning is made) and subsequent follow-ups.

SECONDARY OUTCOMES:
Truncal balance changes | Baseline, then 6-months, 12-months and 24-months follow-ups
  Changes over time between the two groups/arms of brace-weaning protocol
Health-related Quality of Life measure | Baseline, then 6-months,12-months and 24 months follow-ups
  The refined Chinese version of the Scoliosis Research Society-22 (SRS-22r) questionnaire
Health-related Quality of Life measure | Baseline, then 6-months,12-months and 24 months follow-ups
  The EuroQol-5 dimension (EQ-5D) utility score

CONTACTS AND LOCATIONS:
Locations (1):
- Jason Pui Yin Cheung, Hong Kong, Please Select An Option Below, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheung PWH, Chan OKO, Wu H, Lai MKL, Wong LPK, Tang S, Cheung JPY. Immediate vs Gradual Brace Weaning Protocols in Adolescent Idiopathic Scoliosis: A Randomized Clinical Trial. JAMA Pediatr. 2024 Jul 1;178(7):657-668. doi: 10.1001/jamapediatrics.2024.1484. PMID 38829664